CLINICAL TRIAL: NCT06049979
Title: Correlation Between Intestinal Blood Flow and Intestinal Dysfunction in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-PUMCH-A-216
Record Dates: First submitted 2023-09-04; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Critically Ill Patients
Keywords: Intestinal Blood Flow; Acute gastrointestinal injury; Critically Ill Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AGI group: critical ill patient with AGIUS score>2
  Interventions: Other: Acute gastrointestinal injury
- non-AGI group: critical ill patient with AGIUS score 0~2

INTERVENTIONS:
Other: Acute gastrointestinal injury — AGIUS score>2
  Groups: AGI group

SUMMARY:
Currently in the field of critical care, altered intestinal blood flow in critically ill patients has been a hot research topic in recent years. However, because the gastrointestinal tract is in the abdominal cavity and the clinic lacks perfusion direct monitoring means, at present, gastrointestinal function indicators are mostly used to guide the clinic, and the treatment is often blind and lagging. Gastrointestinal perfusion Research on gastrointestinal perfusion is mostly confined to abdominal perfusion pressure (mean arterial pressure - intra-abdominal pressure). However, according to the "Darcy law" in blood flow mechanics, Q=MAP/SVR, which means pressure≠flow. The investigators may not be able to ensure adequate blood flow to the digestive organs by relying on intra-abdominal perfusion pressure alone. Direct organ flow monitoring is a more accurate means of organization.

The superior mesenteric artery (SMA) supplies all of the intestinal tract (small bowel, part of the colon) and is a long vessel that can to reflect the perfusion status of the distal overall bowel. Color Doppler ultrasonography is used to evaluate intestinal vessels such as the SMA in healthy and outpatient patients.

The use of color Doppler ultrasonography to assess blood flow in intestinal vessels such as the SMA in healthy and outpatient patients has been in use since the 1980s. The investigators' team showed that the resistance index of the SMA in postoperative cardiac surgery patients correlated with lactate values and lactate clearance [Front Med (Lausanne), 2021.8:p.762376.], suggesting that gastrointestinal perfusion as reflected by SMA blood flow is important for systemic resuscitation, and that Doppler indices of SMA have the potential value of reflecting intestinal hypoperfusion.

The Doppler index of SMA has the potential value of reflecting intestinal hypoperfusion. Intestinal venous blood enters the portal vein and then the liver before returning to the right heart via the inferior vena cava. Right heart dysfuction, right atrial hypertension, and abdominal hypertension can cause obstruction of portal venous return, which can lead to edema and dysfunction of the bowel. This can lead to edema of the intestinal tract and dysfunction. Therefore, monitoring the venous return status of portal vein, hepatic vein and inferior vena cava is also important for the perfusion of the intestine.

Therefore, monitoring the status of venous return in the portal vein, hepatic vein, inferior vena cava, etc. is also important for intestinal perfusion.

Doppler ultrasound technology has been widely used in the field of cardiac critical care and craniocerebral critical care, but it is still in the exploratory stage in the field of critical care digestion, and this study is an innovative and exploratory one.

DETAILED DESCRIPTION:
Research Methods

(1) Doppler ultrasound technique for intestinal blood flow assessment:An ultrasound system (X-Porte Ultrasound System, FUJIFILM SONOSITE, INC., USA) consisting of a 2-5 MHz C60xp probe was performed. Blood flow parameters were measured by two ICU physicians and the mean values were recorded. Both ICU physicians had more than 4 years of experience in critical care ultrasound; they were certified by the Chinese Critical Care Ultrasound Study Group. SMA flow was measured 1 cm proximal to the abdominal aorta. The insertion angle was <60° . The vessel cross-section was circular. The probe was rotated 90° where the vessel flow was measured and the diameter of the lumen (D) was measured. To minimize errors, it is important to take the average of three measurements in a magnified state. The cross-sectional area of the artery is calculated. Peak systolic velocity (PSV), end-diastolic velocity (EDV), resistance index (RI), time-averaged mean velocity (TAMV), pulsatility index (PI), and blood flow (BF, mL/min) were measured using time-velocity waveform readings according to the calculation software carried by the sonographer. BF=π(D/2)²×TAMV×60, PI=(PSV-EDV)/TAMV, RI=(PSV-EDV)/PSV.

2) Ultrasound score of transabdominal bowel function (AGUIS score) At the time of the ultrasound examination, the operator categorized the situation as "good quality", "poor quality" or "not assessable". The operator categorizes the situation as "good quality," "poor quality," or "not evaluable. The abdomen is then divided into four quadrants, each measuring one point, and the operator examines and scores the diameter of the bowel, changes in bowel folds (e.g., shortening, decreasing), thickness of the bowel wall, layering of the bowel wall, peristalsis, and movement of bowel contents. A total of four scores are obtained, and the average of the four measurements is the (AGIUS) score.

(3) Serologic indices of intestinal mucosal epithelial injury Plasma citrulline, plasma intestinal fatty acid binding protein, and D-lactic acid were measured by ELISA. (R&D Systems, Minneapolis, USA). Peripheral blood specimens were obtained and centrifuged, and the resulting plasma was frozen at -20°C and sent to the laboratory for analysis within 1 week.

Study Route:

Patients with sepsis who met the inclusion criteria were enrolled on the day of enrollment to improve the recording of hemodynamic parameters, measurement of Doppler parameters of intestinal blood flow, and serum specimen retention. Measurements of the above parameters were repeated daily from the first to the third day.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sepsis with an expected ICU stay of more than 3 days.
2. ≥18 years of age and <80 years of age.

Exclusion Criteria:

1. Coronary heart disease, severe mesenteric or abdominal artery stenosis;
2. Fixed body (such as recent spinal surgery or intracranial hypertension);
3. Patients with contraindications for IAP measurement (such as patients who have recently undergone bladder surgery, been injured, or become pregnant;
4. Having undergone abdominal surgery or chest lowering involving the intestines patients undergoing aortic surgery;
5. Poor quality of abdominal ultrasound images;
6. Hydrothorax or ascites.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU admitted patients in comprehensive hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal Ultrasound Score (AGIUS) | Day 1，Day 2，Day 3
  Quantitative scoring is performed by using ultrasound to evaluate intestinal diameter, intestinal wall thickness, and motility. The range is 0-6 points. 0 is the best, 6 is the worst
pulsatile index of superior mesenteric artery | Day 1，Day 2，Day 3
  pulsatile index of superior mesenteric artery

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment（SOFA） | Day 1，Day 2，Day 3
  Sequential Organ Failure Assessment
Mechanical ventilation duration | Total time left from ICU or within 28 days
  Mechanical ventilation duration
28 day mortality rate | Within 28 days after ICU admission
  28 day mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Chair — PUMCH
Locations (1):
- Department of Critical Care Medicine of pekin union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No